CLINICAL TRIAL: NCT02652312
Title: Effect of Dexmedetomidine Infusion on Desflurane Consumption and Hemodynamics During BIS Guided Laparoscopic Surgery: A Randomized Controlled Study
Brief Title: Dexmedetomidine and Desflurane Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Yasser Mostafa Samhan, Professor of Anesthesia, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anesthesia 110T
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
Keywords: Dexmedetomidine; Desflurane; Bispectral Index BIS
MeSH Terms: interventions — Dexmedetomidine; Placebo Effect; Ondansetron; Fentanyl; Propofol; Atracurium; Diclofenac; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 'D' (Active Comparator): Dexmedetomidine group Patients received dexmedetomidine (2 ml diluted in 18 ml of saline) IV in a dose of 1 mcg/kg over 10 minutes. A maintenance dose of Dexmedetomidine infusion at 0.5 mcg/kg/hour was infused.
  Ondansetron: 0.15 mg/kg intravenous preoperative. Fentanyl: 1.5 μg/kg intraoperative Propofol: 10 mg every 5 seconds until the BIS level dropped below 60 for induction of anesthesia.
  Atracurium: 0.5 mg/kg IV. Desflurane: 1 MAC concentration. Diclofenac sodium: 1 mg/kg for postoperative analgesia.
  Interventions: Drug: Dexmedetomidine; Procedure: Ondansetron; Procedure: fentanyl; Procedure: propofol; Procedure: Atracurium; Procedure: diclofenac sodium; Procedure: desflurane
- Group 'P' (Placebo Comparator): Placebo group Patients received similar volume of normal saline as the bolus and maintenance infusion as group D.
  Ondansetron: 0.15 mg/kg intravenous preoperative. Fentanyl: 1.5 μg/kg intraoperative Propofol: 10 mg every 5 seconds until the BIS level dropped below 60 for induction of anesthesia.
  Atracurium: 0.5 mg/kg IV. Desflurane: 1 MAC concentration. Diclofenac sodium: 1 mg/kg for postoperative analgesia.
  Interventions: Drug: Placebo; Procedure: Ondansetron; Procedure: fentanyl; Procedure: propofol; Procedure: Atracurium; Procedure: diclofenac sodium; Procedure: desflurane

INTERVENTIONS:
Drug: Dexmedetomidine — A maintenance dose of Dexmedetomidine infusion at 0.5 mcg/kg/hour made to 20 mL with normal saline will be administered
  Other Names: Precedex; Dexdor
  Arms: Group 'D'
Drug: Placebo — A maintenance dose of 20 mL with normal saline will be administered at a rate similar to that of dexmedetomidine
  Other Names: placebo effect
  Arms: Group 'P'
Procedure: Ondansetron — 0.15 mg/kg intravenous (IV) will be given as a pre-medication
  Other Names: Zofran
Procedure: fentanyl — 1.5 μg/kg intraoperative
  Other Names: Sublimaze,Actiq, Durogesic, Duragesic
Procedure: propofol — 10 mg every 5 seconds until the BIS level dropped below 60 for induction of anesthesia
  Other Names: Diprivan
Procedure: Atracurium — 0.5 mg/kg IV for endotracheal intubation
  Other Names: Atracurium besilate
Procedure: diclofenac sodium — 1 mg/kg for postoperative analgesia
  Other Names: Voltaren
Procedure: desflurane — 1 MAC concentration (expired fraction of 6.0 vol%) for maintenance of anesthesia
  Other Names: Suprane

SUMMARY:
The aim of this study is to calculate desflurane consumption when combined with intraoperative dexmedetomidine infusion guided by bispectral index (BIS)

DETAILED DESCRIPTION:
Forty patients will be randomly allocated into two equal groups as Group 'D' (Dexmedetomidine group) and Group 'P' (Placebo group) using computer generated random numbers. After arrival in the operating room, ondansetron 0.15 mg/kg intravenous (IV) will be given as a pre-medication. Ringer's acetate solution (500 ml) will be infused as a preload then at a rate of 6-8 ml/kg/h during surgery for supplying maintenance and deficit. Monitoring consisted of continuous electrocardiogram (EKG), non-invasive blood pressure (NIBP), pulse oximetry (SpO2), CO2 expired fraction (ETCO2), desflurane inspired fraction (FIdes), and desflurane expired fraction (ETdes) (Infinity Kappa, Dräger, Lübeck, Germany) will be attached to the patient. BIS module (InfinityR BISxTM SmartPodR, smoothing rate: 15 or 30 seconds, software revision: VF5) will also be attached for detection of consciousness level.

All patients will be preoxygenated with 100% oxygen for 3 minutes. The patients in group D will receive dexmedetomidine (2 ml diluted in 18 ml of saline) IV in a dose of 1 mcg/kg over10 minutes through infusion pump prior to induction. Group P patients will receive similar volume of normal saline over 10 min. The study drug and placebo infusions will be prepared by an anesthesiologist who is not involved in the study and the anesthesiologist recording the details is unaware of the type of infusion patients received. Anesthesia will be induced with IV fentanyl 1.5 μg/kg and propofol in a dose of 10 mg every 5 seconds until the BIS level dropped below 60 and confirmed with loss of response to verbal commands. In both groups, Atracurium 0.5 mg/kg IV will be administered, and trachea will be intubated. Fresh gas flow oxygen in air 30-40% at a rate of 3 L/min for 10 minutes will be administered then the flow will be decreased at a rate of 1 L/min using a closed system (Fabius GS, Dräger, Lübeck, Germany) and ventilation will be adjusted to maintain end-tidal carbon dioxide at 30-35 mmHg. Patients in study groups will receive the volatile agent at a concentration of 1 MAC (Minimum Alveolar Concentration). The MAC of desflurane is defined as an expired fraction of 6.0 vol%. Then the dial-up desflurane percentage will be adjusted to establish a BIS value between 40- 50. A maintenance dose of Dexmedetomidine infusion at 0.5 mcg/kg/hour made to 20 mL with normal saline will be administered in group D patients and a similar volume of normal saline will be administered in Group P, till the end of surgery. Top up doses of Atracurium will be given as needed. When heart rate and blood pressure exceeds 20% of baseline in spite of adequate level of anesthesia guided by BIS, boluses of 0.5 μg/kg will be given. While decrease in heart rate and blood pressure more than 20% of baseline, will be treated by ephedrine 5 mg.

In both groups, dexmedetomidine or saline will be stopped approximately 15-20 minutes before completion of surgery, diclofenac sodium 1 mg/kg will be given IM at the time of skin closure. Desflurane will be discontinued after skin closure in both groups. Reversal of neuromuscular blockade will be achieved with neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Tracheal extubation will be done when respiration is satisfactory and adequate muscle tone is achieved

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status of I and II
* undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* history of psychiatric/neurological illness
* cardiovascular disease
* morbid obese patients
* pregnant and nursing women
* known allergic reaction to any of the study medication
* recent use of sedatives or analgesics

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
desflurane consumption (ml) | Intraoperative
  Calculation of desflurane consumption during the intraoperative period

SECONDARY OUTCOMES:
Heart Rate (Beat/min) | Intraoperative
  Recording of the heart rate during the intraoperative period before induction, after induction, after intubation, and then at 5, 10, 15, 30, 45, and 60 minute after intubation and at extubation.
Blood Pressure (mm Hg) | Intraoperative
  Recording of the heart rate during the intraoperative period before induction, after induction, after intubation, and then at 5, 10, 15, 30, 45, and 60 minute after intubation and at extubation.
Fentanyl consumption (ug) | Intraoperative
  Total intraoperative fentanyl consumption

CONTACTS AND LOCATIONS:
Overall Officials: Abla El Hadidy, PhD, Study Director — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harsoor SS, Rani DD, Lathashree S, Nethra SS, Sudheesh K. Effect of intraoperative Dexmedetomidine infusion on Sevoflurane requirement and blood glucose levels during entropy-guided general anesthesia. J Anaesthesiol Clin Pharmacol. 2014 Jan;30(1):25-30. doi: 10.4103/0970-9185.125693. PMID 24574589
- [Background] Kamibayashi T, Maze M. Clinical uses of alpha2 -adrenergic agonists. Anesthesiology. 2000 Nov;93(5):1345-9. doi: 10.1097/00000542-200011000-00030. No abstract available. PMID 11046225
- [Background] Nishibe S, Imanishi H, Mieda T, Tsujita M. The effects of dexmedetomidine administration on the pulmonary artery pressure and the transpulmonary pressure gradient after the bidirectional superior cavopulmonary shunt. Pediatr Cardiol. 2015 Jan;36(1):151-7. doi: 10.1007/s00246-014-0979-2. Epub 2014 Aug 12. PMID 25113519